CLINICAL TRIAL: NCT02863497
Title: The Mindfulness, Incontinence and Sexual Function Treatment Study
Acronym: MIST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment was unfeasible due to patients being unavailable to recruit.
Sponsor: University of British Columbia (Other)
Collaborators: Sexual Medicine Society of North America (Unknown)
Responsible Party: Principal Investigator, Geoffrey Cundiff, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H16-00719
Record Dates: First submitted 2016-08-02; First posted 2016-08-11 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Urinary Incontinence; Sexual Dysfunction
MeSH Terms: conditions — Urinary Incontinence; Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Intervention (Active Comparator): For those randomly selected to receive mindfulness-based sex therapy, they will be asked to participate in four sessions of group therapy, over a period of 2 months. Sessions will occur in a conference room at St. Paul's Hospital. Part of the protocol of the Mindfulness - based sex therapy is that they will have a diary to be filled in. This diary will not be collected at the end of the therapy, as it is for the participant to keep. The group facilitators will be collecting session attendance.
  Interventions: Behavioral: Mindfulness-based Sex Therapy
- No Intervention (No Intervention): For those who are not in the intervention group they will simply be asked to fill the initial questionnaire and the 3 month post questionnaire. They will not participate in any other questionnaires.

INTERVENTIONS:
Behavioral: Mindfulness-based Sex Therapy — These group sessions will include education about sexuality, and the practice of mindfulness skills (including paying attention to the present moment, and to body sensations). Each group will include 7-8 women, plus the group facilitators. The group facilitators for the study will include Dr. Laurel Paterson (who has extensive experience in administering Mindfulness-based sex therapy in other populations of women), and occasionally one of the research team members.
  Arms: Mindfulness Intervention

SUMMARY:
This study aims to determine if there is an impact on sexual distress using mindfulness-based sex therapy (MBST) in addition to standard urogynecologic care, in women with both urinary incontinence (UI) and sexual dysfunction.

DETAILED DESCRIPTION:
Purpose: To evaluate the feasibility of a large multicenter randomized controlled trial to determine the impact on sexual distress of mindfulness-based sex therapy (MBST) in addition to standard urogynecologic care, in women with both urinary incontinence (UI) and sexual dysfunction.

Hypothesis: The addition of MBST to standard urogynecologic care reduces sexual distress in women with UI and sexual dysfunction.

Background/Justification: Sexual dysfunction is a common finding in women over the age of 40 seeking gynecologic care, with 66% of women reporting at least one complaint, and 26% reporting sexual distress. This can have profound negative consequences on health related quality of life, interpersonal relationships, stress level, and mood. Some studies have also shown that the prevalence of sexual dysfunction increases with age, with as many as 80% of elderly women reporting dysfunction. In parallel, urinary incontinence, the involuntary leakage of urine, is also increasingly prevalent with age, with 30-50% of elderly women being affected. Limited evidence suggests that treatments for urinary incontinence, whether conservative or surgical, can improve sexual function. Specifically, after surgery for stress urinary incontinence, 32% of women show improved sexual function, 55% see no change, and 13% report worsened function. Mindfulness is a type of meditation that brings the individual's awareness to the present moment in a non-judgmental manner. Since the 1970s, mindfulness-based therapies have been used increasingly to treat multiple conditions including chronic pain, anxiety, depression, and many others. Mindfulness-based sex therapy (MBST) has been shown to be effective in managing sexual dysfunctions in women with arousal disorders, vulvar pain, a history of gynecological cancer, and a history of sexual abuse. The International Consultation on Sexual Medicine, at the last meeting in June 2015, has recommended the use of mindfulness-based therapy in women with low sexual desire. Mechanisms through which mindfulness is believed to impact sexual function are numerous. First, mindfulness practice produces changes in brain structure and functioning in areas involved in attention, emotion and self-awareness. It also leads to improvements in mood, and decreases stress and anxiety, all of which are major contributors to sexual dysfunction. Second, mindfulness' emphasis on non-judgment can help foster acceptance of the partner. It can also reduce self-criticism associated with a distorted body image. Additionally, improved attention on sensual stimuli and lessened distractibility can increase arousal.

Research Design:

This will be a pilot randomized study of women with UI referred to the Centre for Pelvic Floor, St. Paul's Hospital, in Vancouver, British Columbia, Canada. Recruitment will begin after obtaining ethics approval for the study. All women referred to the Centre for Pelvic Floor complete an intake questionnaire prior to their first consultation. That questionnaire includes a sexual function assessment. Women with identified sexual dysfunction with distress, on baseline questionnaire, will be invited to participate in the proposed study. Potential participants will be first informed about the study by the physician seeing the patient in consultation. If patients are willing to meet the research team, the research coordinator or a trained medical student will further explain the study, and enroll interested women who meet the inclusion and exclusion criteria, while obtaining informed consent to participate. After having completed baseline assessments, participants will then be randomized to the standard urogynecological care control group, or the standard care plus mindfulness-based sex therapy (MBST) intervention group (60 total participants, 30 in each group). Standard urogynecological care for UI varies based on the type of UI and patient preferences, but can include pelvic floor exercises, pelvic floor physiotherapy, medications for bladder function, pessary fitting (a silicone ring placed in the vagina to reduce symptoms of urinary incontinence, as well as pelvic organ prolapse), and/or surgery.

Baseline information will be collected and it will include: participants' demographic characteristics, pelvic floor dysfunction (PFD) and urinary incontinence symptoms, and exam findings, from their first consultation visit assessment. Further information will be obtained with additional questionnaires about body image, mindfulness, anxiety, and depression symptoms.

Women will then undergo management of their UI with or without MBST sessions. Intervention participants (those who undergo MBST session) will then be re-evaluated with the same questionnaires within 2-4 weeks after intervention. All patients will then have their final assessment three months after intervention (including three months post-operatively, to allow time to resume intercourse after the initial surgical healing time).

Data will be collected from patients' charts about their urogynecological management (treatment with pelvic floor exercises, pelvic floor physiotherapy, reduction of dietary triggers, bladder retraining, medications, incontinence pessary, surgery, etc.) as well as their response to treatment.

Throughout the process, the recruitment rates, research coordinator time, methodological barriers, MBST session attendance, and follow-up will all be documented.

Information gathered from this pilot study will inform a future multicenter trial. There is a plan to then disseminate the findings to the medical community involved in women's health, as well as to share them with the public at large.

Statistical Analysis:

Descriptive statistics of demographic characteristics will be included. Pre and post therapy sexual distress will be evaluated and compared between the groups who undergo standard urogynecologic care only vs. standard care plus MBST, with an intention- to-treat analysis. Linear regression on the post therapy score adjusted for pre therapy score on the FSDS-R sexual distress questionnaire will be performed. Standard deviation around the observed difference between the groups will contribute to sample size calculation for a future randomized trial. Secondary pilot outcomes will be descriptively assessed. Secondary trial outcomes will be compared between groups using paired t-test, Wilcoxon rank sum test or linear regression as appropriate. Interaction between treatment and other variables (i.e., severity of UI symptoms at baseline, cure of UI, other PFD symptoms) on sexual function will be assessed using linear regression analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Women 19 years and older with both UI and sexual dysfunction, seen at the Centre for Pelvic Floor, and are interested and available to participate in the study.
2. UI is defined as one of the items below:

   * Stress UI: involuntary loss of urine with increased intra-abdominal pressure (effort, coughing, laughing, sneezing, physical exercise, etc.)

     * Symptoms and positive response to question # 17 of Pelvic Floor Distress Inventory (PFDI-20)
     * Or Positive cough stress test on exam
     * Or positive urodynamics stress UI Urgency UI (also referred to as overactive bladder): involuntary loss of urine with urgency
     * Symptoms and positive response to question # 16 of PFDI-20
     * Or positive urodynamics overactive bladder
   * Mixed UI: combination of stress and urgency UI
   * +/- prolapse or other PFDs concomitantly
   * Can chose any treatment for their condition that is offered to them, but for analysis purposes, must agree to using only one line of treatment during the course of study (should not change treatment during study)
3. Female sexual dysfunctions are categorized by the DSM-5 as sexual interest/arousal disorder, genitopelvic pain/penetration disorder, and female orgasmic disorder. The diagnoses require symptoms to be present for six months or more, for significant distress to be experienced as a result, and for the condition to not be better explained by a mental or medical condition.
4. Sexual distress will be diagnosed as score of 11 or higher on the female sexual dysfunction scale

Exclusion Criteria:

1. Non-English speaking
2. Pregnancy
3. Neurological conditions explaining UI
4. Congenital genitourinary defects
5. Genital fistulas

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-04; Primary Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Improvement in Female Sexual Distress | 3 months post treatment
  To determine the difference in score improvement on the Female Sexual Distress Scale (FSDS-R) between MBST intervention vs. control groups at three months post-treatment

SECONDARY OUTCOMES:
Patient Demographics | 3 month post treatment
  To assess patient retention and treatment response based on demographic characteristics
Patient retention | The study recruitment on average of 1 year
  To recruit a minimum of six women per month
Measuring patient follow up post treatment | 3 months post treatment
  To achieve 80% follow-up at three months post treatment
Sexual Intercourse resumption as assessed by questionnaire | 3 months post treatment
  To observe 75% resumption of sexual intercourse after surgery, in sexually active patients
To collect feedback about the treatment experience through an informal questionnaire | 3 months post treatment
  To obtain informal patient feedback about their involvement
Research coordinator time documentations | From Recruitment to 3 Months Post Treatment
  To document research coordinator time needed per participant in this population of generally older women (compared to existing studies on MBST)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey W. Cundiff, Principal Investigator — UBC Obstetrics & Gynaecology; Maryse Larouche, Principal Investigator — Obstetrics & Gynaecology; Lori Brotto, Principal Investigator — UBC Obstetrics & Gynaecology
Locations (1):
- Centre for Pelvic Floor, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No